CLINICAL TRIAL: NCT05403476
Title: A Randomised, Double-blind, Placebo-controlled Trial to Assess the Efficacy and Safety of FE 999049 for Treatment of Men With Idiopathic Infertility
Brief Title: A Trial to Compare Efficacy and Safety of Follitropin Delta Versus Placebo (Inactive Treatment) in the Treatment of Men With Idiopathic Infertility (Unexplained Reduction of Semen Quality) (ADAM)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The probability of enrolling subjects in the trial in a reasonable timeframe was too low. The termination was not due to safety concerns nor changes in Ferring's Reproductive Medicine strategy or interest in developing treatments for Male Infertility
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000400
Record Dates: First submitted 2022-05-30; First posted 2022-06-03 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-08

CONDITIONS: Male Idiopathic Infertility
MeSH Terms: interventions — FE 999049; follitropin delta

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FE 999049 (Follitropin Delta) (Experimental)
  Interventions: Drug: FE 999049
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FE 999049 — FE 999049 is administered as single daily subcutaneous injections of 12 μg for 6 months.
  Other Names: REKOVELLE; Follitropin Delta
  Arms: FE 999049 (Follitropin Delta)
Drug: Placebo — Placebo is administered as single daily subcutaneous injection dialed to the same value (dose) as FE 999049 for 6 months.
  Arms: Placebo

SUMMARY:
The primary purpose of this trial is to investigate whether men with idiopathic infertility (unexplained reduction of semen quality), after being treated with a daily dose of 12 µg recombinant follicle stimulating hormone (rFSH) for 6 months, can improve the chance of spontaneous pregnancy observed in their female partners in comparison to placebo (inactive treatment). For more information, please visit the trial's website www.adamclinicaltrial.com (only applicable in the US).

ELIGIBILITY:
Inclusion Criteria:

* History of infertility with current partner at randomisation must be 12-60 months if current partner is aged <35 years or 6-60 months if current partner is aged 35-38 years.
* Men between the ages of 18 and 50 years.
* Total sperm count 5-39 million at screening; confirmed by two consecutive samples taken ≥2 weeks apart before randomization.
* Total sperm motility of ≥10% at screening; confirmed by two samples taken ≥2 weeks apart before randomisation. If a semen sample has been taken within 3 months prior to screening and been analysed at an andrology laboratory, it can be included as the first of the two semen samples at screening.
* Semen volume ≥1.4 mL at screening; confirmed by two consecutive samples taken ≥2 weeks apart before randomization.
* Serum follicle-stimulating hormone (FSH) levels of 2-12.0 IU/L (measured at central laboratory) at screening)
* Serum luteinising hormone (LH) levels of 1.2-7.5 IU/L (measured at central laboratory) at screening.
* Serum total testosterone levels of ≥300 ng/dL (equals ≥10.4 nmol/L; measured at central laboratory) at screening.
* Agree to have regular intercourse with current female partner with the intent of spontaneous conception within 9 months from randomization.
* Agree to provide information on female partner's positive urine pregnancy test(s) and documentation of ultrasound(s), delivery, and neonatal/infant health.

Current partner fulfilling the criteria below:

* Pre-menopausal woman between the ages of 18 and 38 years (both inclusive) at the time of randomisation of male participant.
* Regular menstrual cycles of 21-35 days.
* No history or current condition of pelvic inflammatory disease, endometriosis stage II-IV by definite or empirical diagnosis, or tubal ligation.
* Agree not to obtain infertility treatment outside of this trial for 6 months from randomization of male subject.

Exclusion Criteria:

* Previous FSH treatment for ≥4 months not leading to conception.
* Past or current use of finasteride within 3 months prior to screening.
* Any history of anatomical disorder of the pituitary gland or testes.
* Any structural abnormalities of the vas deferens (unilateral or bilateral) at screening.
* Any known, clinically significant, systemic disease in addition to the trial indication that might negatively impact fertility.
* Known history or presence of clinical varicocele (subclinical and Grade 1 varicocele are acceptable).
* Known history of cryptorchidism, testicular torsion, or orchitis.
* Known abnormal karyotype (including Y-chromosome microdeletion).
* Current or past treatment of urogenital (kidney, bladder, testicular, or prostate) cancer as well as history of chemo- or radiotherapy that can have impact on testes.
* Any known uncontrolled non-gonadal endocrinopathies (thyroid, adrenal, pituitary disorders).
* Administration of hormonal preparations, agents known to impair testicular function or affect sex hormone secretion, and known or suspected teratogens within 3 months prior to screening. Administration of anabolic steroids within 12 months prior to screening.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 4 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2024-10-05 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Spontaneous pregnancy observed in female partner within 9 months after randomization of male subject, where spontaneous pregnancy is defined as vital pregnancy | Up to 9 months after randomization
  Vital pregnancy is documentation of at least one intrauterine gestational sac with fetal heartbeat by ultrasound.

SECONDARY OUTCOMES:
Positive Beta-Human Chorionic Gonadotropins (βhCG) (positive urine βhCG test) observed in female partner | Up to 9 months (End-of-Trial)
Time from randomization to spontaneous pregnancy observed in female partner in calendar time and number of menstrual cycles | Up to 9 months (End-of-Trial)
Changes in semen volume from pre-randomization to 3, 6, and 9 months after randomization | From pre-randomization to 3, 6 and 9 months after randomization
Changes in sperm concentration from pre-randomization to 3, 6, and 9 months after randomization | From pre-randomization to 3, 6 and 9 months after randomization
Changes in total sperm count from pre-randomization to 3, 6, and 9 months after randomization | From pre-randomization to 3, 6 and 9 months after randomization
Changes in total motile sperm count from pre-randomization to 3, 6, and 9 months after randomization | From pre-randomization to 3, 6 and 9 months after randomization
Changes in sperm morphology from pre-randomization to 3, 6, and 9 months after randomization | From pre-randomization to 3, 6 and 9 months after randomization
Changes in semen DNA fragmentation from pre-randomization to 3, 6, and 9 months after randomization | From pre-randomization to 3, 6 and 9 months after randomization
Treatment responders defined by either spontaneous pregnancy observed in female partner, or increase of total sperm count or total motile sperm count to 50% over average baseline at 6 and/or 9 months | Baseline to 6 and 9 months
Changes in follicle stimulating hormone (FSH) from randomization to 3 and 6 months after randomization | From randomization to 3 and 6 months after randomization
Changes in luteinising hormone (LH) from randomization to 3 and 6 months after randomization | From randomization to 3 and 6 months after randomization
Changes in inhibin B from randomization to 3 and 6 months after randomization | From randomization to 3 and 6 months after randomization
Changes in testosterone from randomization to 3 and 6 months after randomization | From randomization to 3 and 6 months after randomization
Changes in estradiol from randomization to 3 and 6 months after randomization | From randomization to 3 and 6 months after randomization
Changes in free testosterone concentration from randomization to 3 and 6 months after randomization | From randomization to 3 and 6 months after randomization
  Blood samples for assessment of sex hormone binding globulin (SHBG) concentrations will be drawn in order to calculate free testosterone concentrations.
Treatment-induced anti-FSH antibodies, overall as well as with neutralising capacity | From randomization to 21-35 days after End-of-treatment
  Blood samples for assessment of anti-FSH antibodies will be drawn.
Immune-related adverse events | From randomization to End-of-Trial (up to 9 months)
  All treatment-emergent adverse events will be analyzed to identify those that potentially are immune related.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (22):
- United States (13):
  - Ferring Investigational Site, Tempe, Arizona
  - Ferring Investigational Site, San Jose, California
  - Ferring Investigational Site, Centennial, Colorado
  - Ferring Investigational Site, Newark, Delaware
  - Ferring Investigational Site, Chicago, Illinois
  - Ferring Investigational Site, Kansas City, Kansas
  - Ferring Investigational Site, New York, New York
  - Ferring Investigational Site, Raleigh, North Carolina
  - Ferring Investigational Site, Oklahoma City, Oklahoma
  - Ferring Investigational Site, Bedford, Texas
  - Ferring investigational site, Webster, Texas
  - Ferring Investigational Site, Salt Lake City, Utah
  - Ferring Investigational Site, Seattle, Washington
- Ferring Investigational Site, Brussels, Belgium
- Ferring Investigational Site, Copenhagen, Denmark
- Germany (2):
  - Ferring Investigational Site, Halle
  - Ferring Investigational Site, Münster
- Italy (2):
  - Ferring Investigational Site, Modena
  - Ferring Investigational Site, Rome
- Ferring Investigational Site, Valencia, Spain
- Sweden (2):
  - Ferring Investigational Site, Malmo
  - Ferring Investigational Site, Stockholm

IPD SHARING:
Plan to Share IPD: No